CLINICAL TRIAL: NCT00910689
Title: Drug and Non-Drug Treatment of Severe Migraine
Acronym: TSM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Merck Sharp & Dohme LLC (Industry); GlaxoSmithKline (Industry)
Responsible Party: Kenneth Holroyd, Distinguished Professor. Department of Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2R01NS032374 (NIH); NS32374
Record Dates: First submitted 2008-11-24; First posted 2009-06-01 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-10

CONDITIONS: Migraine Headache
Keywords: Migraine Headache; Preventive Therapy; Beta Blocker Medication; Behavior Therapy; Clinical Trial
MeSH Terms: conditions — Migraine Disorders | interventions — Propranolol; Nadolol; Behavior Therapy; Sumatriptan; rizatriptan; Metoclopramide; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Optimal Acute Therapy plus Beta Blocker Placebo
  Interventions: Drug: Placebo control; Drug: Optimal Acute Therapy
- 2 (Active Comparator): Optimal Acute Therapy plus Beta Blocker (propranolol or nadolol)
  Interventions: Drug: Propranolol or nadolol; Drug: Optimal Acute Therapy
- 3 (Active Comparator): Optimal Acute Therapy plus Behavioral Migraine Management plus Beta Blocker placebo
  Interventions: Drug: Placebo control; Behavioral: Behavioral Migraine Management (BMM); Drug: Optimal Acute Therapy
- 4 (Active Comparator): Optimal Acute Therapy plus Behavioral Migraine Management plus Beta Blocker (propranolol or nadolol)
  Interventions: Drug: Propranolol or nadolol; Behavioral: Behavioral Migraine Management (BMM); Drug: Optimal Acute Therapy

INTERVENTIONS:
Drug: Propranolol or nadolol — Treatment initiated with 1 capsule (60 mg long acting propranolol hydrochloride) and increased to 3 capsules (180 mg) at week 12 as tolerated. If subject does not tolerate at least 2 capsules (120 mg) of propranolol hydrochloride-LA, and in treating neurologist's judgment are unimproved, subject switched to second medication (nadolol). Participants initially receive a single 40 mg capsule of nadolol and increased to 2 capsules (80 mg) as tolerated. At week 12 dose stabilized at highest tolerated level. In evaluation phase, an increase to 4 capsules of long acting propranolol hydrochloride (240 mg) or 3 capsules of nadolol (120 mg) permitted.
  Other Names: Inderal; Nadolol
  Arms: 2; 4
Drug: Placebo control — Placebo
  Arms: 1; 3
Behavioral: Behavioral Migraine Management (BMM) — Session 1: Overview of the pathophysiology of migraine; introduce muscle stretching, deep breathing, PMR, imagery; Session 2: Development trigger management strategy; Use early warning signs as a cue to use behavioral migraine management and acute medication; Session 3:(a) continue with "basic" migraine management skills if these skills have not been mastered;(b) introduce cognitive-behavioral stress-management, if stress is a salient migraine trigger;(c) introduce thermal biofeedback ("hand warming") training with a portable home thermal biofeedback device, if stress is not a notable migraine trigger. Session 4: Review problems using various behavioral migraine management skills; Prepare written migraine management plan; Relapse prevention addressed
  Other Names: Behavioral Treatment; BMM
  Arms: 3; 4
Drug: Optimal Acute Therapy — This acute therapy protocol emphasized treatment with a 5-HT1B/D-agonist or triptan. Nonsteroidal anti-inflammatory (NSAID; ibuprofen) and anti-emetic (metoclopramide) medication could be added as needed. The choice of triptans (rizatriptan®, sumatriptan®), the route(s) of triptan administration (oral, nasal spray, subcutaneous injection), and the addition of a NSAID, or anti-emetic were tailored to participant preference, treatment history and acute therapy response. Individualized handouts and a phone call (week 3) of the OAT Run-in were used to help participants evaluate and optimize their acute therapy.
  Other Names: Imitrex®; Maxalt®; Reglan®; Advil®; Motrin®; Nuprin®

SUMMARY:
The purpose of this study is to determine if the addition of preventive medication, behavior migraine management or the combination of preventive medication and behavior migraine management improves the outcome of optimal acute therapy for frequent migraines.

DETAILED DESCRIPTION:
During the 5 week Optimal Acute Therapy (OAT) Run in (Month 1) all participants who met initial inclusion criteria received "optimal" acute therapy (OAT). At the end of the OAT Run-in, participants who continued to meet the migraine severity criteria were stratified by sex and randomized via a computerized randomization procedure to the four added treatments: Beta Blocker Placebo (PL), Beta Blocker (Propranolol LA or Nadolol), Behavioral Migraine Management (BMM) + PL, or BMM + Beta Blocker. Each of the 4 treatment protocols required 4 monthly clinic visits and 3 telephone contacts during the 3 month Treatment/Dose Adjustment Phase (Month 2 to Month 4) where Beta Blocker or PL dose was adjusted and BMM was administered. During the 12 month (Month 5 to Month 16) Evaluation Phase clinic visits were scheduled at Month 5, Month 7, Month 10 (the Primary End Point), Month 13 and Month 16. Treatment conditions were blinded only for the preventive medication (Beta Blocker, Placebo) component, and not for the administration of BMM. Electronic headache diary recordings are obtained for the full 16 months of the trial, including the 12 month evaluation phase, and migraine-related impairments in quality of life are assessed at multiple points over the 16 months of the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years
* Diagnosis of migraine with or without aura (International Classification of Headache Disorders)
* 3 or more migraine episodes/month with disability for the past 6 months
* Less than 20 total headache days/month for the past 6 months

Exclusion Criteria:

* Medication overuse headaches
* Currently taking medications contraindicated by study protocol and unable or unwilling to withdraw
* Concurrently undergoing counseling/psychotherapy treatment
* Unable to read, understand or record information in study diaries, questionnaires, and migraine management manual.
* Unable/unwilling to give written informed consent
* History of exclusionary medical condition such as, but not limited to, epilepsy, heart disease, kidney disease, liver disease, hepatic or renal impairment, stroke, ischemic abdominal syndromes, peripheral vascular disease.
* Uncontrolled hypertension at screening (sitting systolic pressure > 160 mmHg, diastolic pressure > 95 mmHg)
* Fertile female who is breastfeeding, pregnant planning a pregnancy within the next year or is unwilling to use adequate contraception.
* Has exclusionary medical condition such as but not limited to diabetes (insulin dependent), tuberculosis, bronchospastic disease (asthma), heart disease (or multiple risk factors for heart disease), angina pectoris, documented silent ischemia, or cardiac arrythmias requiring medication, or a clinically significant EKG abnormality.
* Other pain diagnosis is primary presenting problem (e.g., fibromyalgia)
* Has a substance abuse problem or a psychological disorder that prevents participation in study (e.g., unmanaged severe depression that requires immediate treatment or limits participation in home-based treatment)
* Hypersensitivity, intolerance or contraindication to use of Propranolol, Nadolol, Sumatriptan, or Rizatriptan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2001-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Holroyd, Ph.D., Principal Investigator — Ohio University
Locations (2):
- United States (2):
  - Ohio University, Athens, Ohio
  - OrthoNeuro, Inc., Westerville, Ohio

REFERENCES:
- [Background] Martin BC, Pathak DS, Sharfman MI, Adelman JU, Taylor F, Kwong WJ, Jhingran P. Validity and reliability of the migraine-specific quality of life questionnaire (MSQ Version 2.1). Headache. 2000 Mar;40(3):204-15. doi: 10.1046/j.1526-4610.2000.00030.x. PMID 10759923
- [Derived] Holroyd KA, Cottrell CK, O'Donnell FJ, Cordingley GE, Drew JB, Carlson BW, Himawan L. Effect of preventive (beta blocker) treatment, behavioural migraine management, or their combination on outcomes of optimised acute treatment in frequent migraine: randomised controlled trial. BMJ. 2010 Sep 29;341:c4871. doi: 10.1136/bmj.c4871. PMID 20880898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient clinics
Pre-assignment Details: 5 week Optimal Acute Therapy (OAT) Run in (M1) precedes random assignment (see detailed design description).
Groups:
- OAT + Placebo (PL): Optimal Acute Therapy plus Beta Blocker Placebo
- OAT + Beta Blocker (Beta-B): Optimal Acute Therapy plus Beta Blocker (propranolol or nadolol)
- OAT + BMM + PL: Optimal Acute Therapy plus Behavioral Migraine Management plus placebo
- OAT + BMM + Beta-B: Optimal Acute Therapy plus Behavioral Migraine Management plus Beta Blocker (propranolol or nadolol)
Period: Month 1: Optimal Acute Therapy Run in
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Started | 55 | 53 | 55 | 69
Completed | 53 | 52 | 50 | 59
Not Completed | 2 | 1 | 5 | 10
Not completed — No Post OAT Run-in data | 2 | 1 | 5 | 10
Period: Month 2- 4: Treatment Period
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Started | 53 | 52 | 50 | 59
Completed | 44 | 42 | 42 | 48
Not Completed | 9 | 10 | 8 | 11
Not completed — Lost to Follow-up | 3 | 4 | 1 | 3
Not completed — Adverse Event | 2 | 3 | 2 | 0
Not completed — Time Demands | 1 | 0 | 4 | 8
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Perceived Improvement | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Period: Months 5 - 10: Evaluation Period I
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Started | 44 | 42 | 42 | 48
Completed | 40 | 35 | 35 | 41
Not Completed | 4 | 7 | 7 | 7
Not completed — Lost to Follow-up | 2 | 5 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 4
Not completed — Lack of Efficacy | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 2 | 0
Not completed — Time Demands | 0 | 0 | 1 | 1
Period: Months 11- 16: Evaluation Period II
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Started | 40 | 35 | 35 | 41
Completed | 30 | 25 | 28 | 35
Not Completed | 10 | 10 | 7 | 6
Not completed — Lost to Follow-up | 3 | 0 | 1 | 2
Not completed — Adverse Event | 2 | 4 | 2 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 3 | 1
Not completed — Time Demands | 2 | 1 | 0 | 0
Not completed — Perceived Improvement | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B | Total
Number analyzed (Participants) | 55 | 53 | 55 | 69 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 53 | 55 | 69 | 232
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.2) | 37.7 (10.1) | 37.1 (9.4) | 38.3 (10.9) | 38.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 45 | 49 | 184
  Male | 10 | 8 | 10 | 20 | 48
Region of Enrollment [Number; unit: participants]
  United States | 55 | 53 | 55 | 69 | 232

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Migraine Episodes Per 30 Days at Month 10.
Description: Change in number of migraine episodes(with 24 hours pain free period required between episodes)per 30 days from OAT run-in (Month 1) to Month 10.Obtained from daily electronic diary.
Time Frame: Change from Month 1 to Month 10
Population: Efficacy analyses were intent-to-treat analyses that included all randomized (N = 232) participants.
Measure: Mean (95% Confidence Interval); unit: Number of Migraine episodes
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Number analyzed (Participants) | 55 | 53 | 55 | 69
Number of Migraine episodes | -2.1 [-2.2 to -1.9] | -2.1 [-2.2 to -1.9] | -2.2 [-2.4 to -2.0] | -3.3 [-3.5 to -3.2]
Statistical Analysis 1: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL vs OAT + BMM + Beta-B; Omnibus Test: A mixed model with fixed effects for treatment,natural time(defined as natural log of months) and treatment-by-time interaction was used to obtain maximum likelihood estimates of missing values and to evaluate treatment effects(using the PROC MIXED procedure in SAS statistical software,version 9;www.sas.com). A significant treatment by time interaction(p < .05, 2-tailed) was followed by post-tests (see below). Details of significant post tests are reported as separate analyses; Test type: Superiority or Other; p < .01, Mixed Models Analysis — Post tests consisted of 6 pair wise contrasts: The first 3 contrasts compared each of the 3 additive treatments (Trial Arms 2, 3, 4) to OAT + PL (Trial arm 1); 3 additional contrasts compared the 3 additive treatments to one another; A Bonferoni procedure was used to control the family-wise type I error for the 6 post test contrasts at .05. Adjusted p =.0083
Statistical Analysis 2: Comparison: OAT + Placebo (PL) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 1.2, Standard Deviation 0.57
Statistical Analysis 3: Comparison: OAT + Placebo (PL) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .25, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 108; Mean Difference (Net) = 0.1, Standard Deviation 0.68
Statistical Analysis 4: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B); Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .98, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.0, Standard Deviation 0.59
Statistical Analysis 5: Comparison: OAT + BMM + PL vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 1.1, Standard Deviation 0.69
Statistical Analysis 6: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 120; Mean Difference (Net) = 1.3, Standard Deviation 0.61
Statistical Analysis 7: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .29, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.1, Standard Deviation 0.72

2. Secondary Outcome: Change in the Number of Migraine Days Per 30 Days at Month 10
Description: Change in the number of days with migraine per 30 days at Month 10 relative to the OAT Run-in (Month 1). Obtained from daily electronic diary.
Time Frame: Change from Month 1 to Month 10
Population: Efficacy analyses were intent-to-treat analyses that included all randomized (N = 232) participants.
Measure: Mean (95% Confidence Interval); unit: Number of days
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Number analyzed (Participants) | 55 | 53 | 55 | 69
Number of days | -3.3 [-3.6 to -3.0] | -3.9 [-4.2 to -3.5] | -3.3 [-3.7 to -2.9] | -5.4 [-5.6 to -5.2]
Statistical Analysis 1: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL vs OAT + BMM + Beta-B; Omnibus test:A mixed model with fixed effects for treatment, time (defined as the natural log of months), and the treatment-by-time interaction was used to obtain maximum likelihood estimates of missing values and to evaluate treatment effects (PROC MIXED, SAS 9).When the treatment by time interaction was significant (p < .05, 2-tailed)post-tests were conducted (see below).Details of significant post tests are reported as separate analyses; Test type: Superiority or Other; p < .03, Mixed Models Analysis — 6 pair wise contrasts were conducted: The first 3 contrasts compared each of the 3 additive treatments to OAT + PL. The 3 additional contrasts compared the 3 additive treatments to one another; A Bonferoni procedure was used to control the family wise type I error for the 6 post test contrasts at .05. Adjusted p =.0083
Statistical Analysis 2: Comparison: OAT + Placebo (PL) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 2.0, Standard Deviation 1.03
Statistical Analysis 3: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 1.5, Standard Deviation 1.12
Statistical Analysis 4: Comparison: OAT + BMM + PL vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 2.1, Standard Deviation 1.26
Statistical Analysis 5: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B); Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .02, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.5, Standard Deviation 1.20
Statistical Analysis 6: Comparison: OAT + Placebo (PL) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .79, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 108; Mean Difference (Net) = 0.1, Standard Deviation 1.35
Statistical Analysis 7: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .02, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Mean Difference (Net) = 0.6, Standard Deviation 1.43

3. Secondary Outcome: Change in Quality of Life at Month 10
Description: Change in Migraine Specific Quality of Life Questionnaire (MSQL; Martin, et al., 2000: v 2.1) scores at Month 10 relative to OAT run-in (Month 1). The MSQL is a 14-item self-report measure that assesses the impact of migraine. The total score ranges from 14 to 84 with higher scores reflecting greater impairment.
Time Frame: Change from Month 1 to Month 10
Population: Efficacy analyses were intent-to-treat analyses that included all randomized (N = 232) participants.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Number analyzed (Participants) | 55 | 53 | 55 | 69
Scores on a scale | -7.1 [-7.8 to -6.3] | -7.1 [-7.7 to -6.6] | -8.6 [-8.9 to -8.2] | -13.0 [-13.5 to -12.5]
Statistical Analysis 1: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL vs OAT + BMM + Beta-B; Omnibus test:A mixed model with fixed effects for treatment, time (defined as the natural log of months), and the treatment-by-time interaction and pretreatment Migraine Specific Quality of Life scores as covariate was used to obtain maximum likelihood estimates of missing values and to evaluate treatment effects (using the PROC MIXED procedure in SAS statistical software, version 9; www. sas.com).A significant treatment by time interaction (p < .05, 2-tailed) was followed by post-tests; Test type: Superiority or Other; p < .005, Mixed Models Analysis — Post tests consisted of 6 pair wise contrasts: The first 3 contrasts compared each of the 3 additive treatments (Trial Arms 2, 3, 4) to OAT + PL (Trial arm 1); three additional contrasts compared the 3 additive treatments to one another; A Bonferoni procedure controlled the familywise type I error for the 6 contrasts at .05. Adjusted p=.0083
Statistical Analysis 2: Comparison: OAT + Placebo (PL) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 108; Mean Difference (Net) = 1.5, Standard Deviation 2.18
Statistical Analysis 3: Comparison: OAT + Placebo (PL) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 6.0, Standard Deviation 2.41
Statistical Analysis 4: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 1.4, Standard Deviation 1.67
Statistical Analysis 5: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 120; Mean Difference (Net) = 5.9, Standard Deviation 2.03
Statistical Analysis 6: Comparison: OAT + BMM + PL vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 4.5, Standard Deviation 1.83
Statistical Analysis 7: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B); Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .87, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.1, Standard Deviation 2.38

4. Secondary Outcome: Change in Number of Migraine Episodes Per 30 Days at Month 16.
Description: Change in number of migraine episodes (with 24 hours pain free period required between episodes) per 30 days from OAT run-in (Month 1) to Month 16. Assessed by participant daily electronic diary.
Time Frame: Change from Month 1 to Month 16
Population: Efficacy analyses were intent-to-treat analyses that included all randomized (N = 232) participants.
Measure: Mean (95% Confidence Interval); unit: Number of Migraine Episodes
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Number analyzed (Participants) | 55 | 53 | 55 | 69
Number of Migraine Episodes | -2.5 [-2.6 to -2.3] | -2.5 [-2.8 to -2.2] | -2.7 [-2.9 to -2.5] | -3.8 [-4.0 to -3.5]
Statistical Analysis 1: Comparison: OAT + Placebo (PL) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 1.3, Standard Deviation 0.77
Statistical Analysis 2: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B); Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .83, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.0, Standard Deviation 0.79
Statistical Analysis 3: Comparison: OAT + Placebo (PL) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .05, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 108; Mean Difference (Net) = 0.2, Standard Deviation 0.67
Statistical Analysis 4: Comparison: OAT + BMM + PL vs OAT + BMM + Beta-B; Significant post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 1.1, Standard Deviation 0.86
Statistical Analysis 5: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 120; Mean Difference (Net) = 1.3, Standard Deviation 0.95
Statistical Analysis 6: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .20, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.2, Standard Deviation 0.89

5. Secondary Outcome: Change in the Number of Migraine Days Per 30 Days at Month 16
Description: Change in the number of migraine days per 30 days at Month 16 relative to the OAT run-in (Month 1). Assessed by participant electronic diary.
Time Frame: Change form Month 1 to Month 16
Population: Efficacy analyses were intent-to-treat analyses that included all randomized (N = 232) participants.
Measure: Mean (95% Confidence Interval); unit: Number of Days
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Number analyzed (Participants) | 55 | 53 | 55 | 69
Number of Days | -3.9 [-4.3 to -3.5] | -4.5 [-5.1 to -4.0] | -4.1 [-4.5 to -3.8] | -6.1 [-6.6 to -5.6]
Statistical Analysis 1: Comparison: OAT + Placebo (PL) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 2.2, Standard Deviation 1.70
Statistical Analysis 2: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 120; Mean Difference (Net) = 1.6, Standard Deviation 1.96
Statistical Analysis 3: Comparison: OAT + BMM + PL vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 2.0, Standard Deviation 1.69
Statistical Analysis 4: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B); Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > .04, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.6, Standard Deviation 1.69
Statistical Analysis 5: Comparison: OAT + Placebo (PL) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > 0.33, t-test, 2 sided — Bonerfoni adjusted critical value p = .0083; Degrees of freedom = 1 and 108; Mean Difference (Net) = 0.2, Standard Deviation 1.34
Statistical Analysis 6: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > 0.21, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.2, Standard Deviation 1.68

6. Secondary Outcome: Change in Quality of Life at Month 16
Description: Change in Migraine Specific Quality of Life Questionnaire (MSQL; Martin, et al., 2000: v 2.1) scores relative to OAT run-in. The MSQL is a 14-item self-report measure that assesses the impact of migraine. The total score ranges from 14 to 84 with higher scores reflecting greater impairment.
Time Frame: Change from Month 1 to Month 16
Population: Efficacy analyses were intent-to-treat analyses that included all randomized (N = 232) participants.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | OAT + Placebo (PL) | OAT + Beta Blocker (Beta-B) | OAT + BMM + PL | OAT + BMM + Beta-B
Number analyzed (Participants) | 55 | 53 | 55 | 69
Scores on a scale | -8.8 [-9.5 to -8.1] | -8.5 [-9.4 to -7.6] | -9.6 [-10.3 to -9.0] | -15.2 [-16.0 to -14.4]
Statistical Analysis 1: Comparison: OAT + Placebo (PL) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 6.4, Standard Deviation 3.00
Statistical Analysis 2: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 6.7, Standard Deviation 3.29
Statistical Analysis 3: Comparison: OAT + BMM + PL vs OAT + BMM + Beta-B; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p < .001, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 122; Mean Difference (Net) = 5.6, Standard Deviation 2.99
Statistical Analysis 4: Comparison: OAT + Placebo (PL) vs OAT + Beta Blocker (Beta-B); Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > 0.56, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 0.3, Standard Deviation 2.85
Statistical Analysis 5: Comparison: OAT + Placebo (PL) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > 0.08, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 108; Mean Difference (Net) = 0.8, Standard Deviation 2.45
Statistical Analysis 6: Comparison: OAT + Beta Blocker (Beta-B) vs OAT + BMM + PL; Post-test contrast. Mean difference in change; Test type: Superiority or Other; p > 0.03, t-test, 2 sided — Bonferoni adjusted critical value p = .0083; Degrees of freedom = 1 and 106; Mean Difference (Net) = 1.1, Standard Deviation 2.83

ADVERSE EVENTS:
Groups:
- OAT + Placebo (PL) at Month 5: Optimal Acute Therapy (OAT) + Beta-Blocker (Propranolol/ Nadolol)Placebo. Side-effects (Fatigue, Gastrointestinal Distress, Insomnia, Lightheaded or Dizzy, Difficulty Concentrating, Depression, Weight Gain, Exercise Intolerance, Nightmares, Drowsiness or Other side effect at Month 5 following dose adjustment.
- OAT + Beta-Blocker at Month 5: Optimal Acute Therapy (OAT) + Beta-Blocker (Propranolol/Nadolol. Side-effects (Fatigue, Gastrointestinal Distress, Insomnia, Lightheaded or Dizzy, Difficulty Concentrating, Depression, Weight Gain, Exercise Intolerance, Nightmares, Drowsiness or other side-effect assessed after dose adjustment(Month 5).
- OAT + BMM + PL at Month 5: Optimal Acute Therapy + Behavioral Migraine Management(BMM) + Beta-Blocker(Propranolol/Nadolol) Placebo.
  Side-effects (Fatigue, Gastrointestinal Distress, Insomnia, Lightheaded or Dizzy, Difficulty Concentrating, Depression, Weight Gain, Exercise Intolerance, Nightmares, Drowsiness or other side-effect)as assessed after dose adjustment(Month 5).
- OAT + BMM + Beta-Blocker at Month 5: Optimal Acute Therapy (OAT)+ Behavioral Migraine Management (BMM)+ Beta-Blocker(Propranolol/Nadolol).
  Side-effects (Fatigue, Gastrointestinal Distress, Insomnia, Lightheaded or Dizzy, Difficulty Concentrating, Depression, Weight Gain, Exercise Intolerance, Nightmares, Drowsiness or other side effect) assessed after dose adjustment(Month 5).
Arm/Group | OAT + Placebo (PL) at Month 5 | OAT + Beta-Blocker at Month 5 | OAT + BMM + PL at Month 5 | OAT + BMM + Beta-Blocker at Month 5
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/53 | 0/55 | 0/69
Other Adverse Events (participants affected / at risk) | 3 | 7 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | OAT + Placebo (PL) at Month 5 | OAT + Beta-Blocker at Month 5 | OAT + BMM + PL at Month 5 | OAT + BMM + Beta-Blocker at Month 5
Fatigue (General disorders) | 3/44 (3) | 7/42 (7) | 2/42 (2) | 2/48 (2)

LIMITATIONS AND CAVEATS:
No side effect reached the 5% reporting threshold at either the Month 10 or the Month 16 assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No